CLINICAL TRIAL: NCT06530264
Title: Evaluation of Different Methods of Posterior Flaps Management in External Dacryocystorhinostomy
Brief Title: Evaluation of Different Methods of Posterior Flap Management in External Dacryocystorhinostomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohammed Sayed Abdelmaaboud Abdelmoneem, Mohammed Sayed Abdelmaaboud, Minia University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Posterior flap managing in DCR
Record Dates: First submitted 2024-07-19; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Acquired Nasolacrimal Duct Obstruction
Keywords: Posterior flap; DCR; NLDO

STUDY DESIGN:
Intervention Model Description: All patients included in this study will be verbally briefed about the details and the nature of the study & will sign a written consent according to the local Ethics Committee of Minia University Faculty of Medicine. The study will be conducted in Ophthalmology department, Minia university Hospital, Egypt.
Masking Description: 1. Patients with chronic dacryocystits,
  2. primary nasolacrimal duct obstruction
  3. Lacrimal mucocele
  4. Lacrimal fistula
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- External DCR (Other): Different techniques in posterior flap management
  Interventions: Other: DCR

INTERVENTIONS:
Other: DCR — 6. An H shaped incision at the postero-inferior lacrimal sac is made, with a long anterior flap and shorter posterior flap. Similarly an H shaped incision at the nasal mucosa is made. The posterior flap of lacrimal sac is sutured with posterior flap of nasal mucosa in interrupted fashion using 6-0 vicryl sutures in Group A, while in Group B the posterior flap is trimmed without suturing.
  Other Names: posterior flap management

SUMMARY:
The aim of DCR is to form a new, mucosa-lined pathway between the lacrimal sac and the nasal cavity where tears can bypass a lacrimal obstruction and drain directly in the nose. The original external approach was described in 19046. In 1920s, mucosal flap anastomosis was added to the procedure as a modification7, and since then, many new modifications have been made to improve the original procedure.

DETAILED DESCRIPTION:
Aim of The Study

• To compare intraoperative details and postoperative endonasal endoscopic findings and their effects on success rate of external dacryocystorhinostomy with and without anastomosis of posterior mucosal flaps.

Patients and Methods

Study Design: This will be a prospective interventional comparative clinical study. It will include two groups according to the surgical procedure:- Group A: includes 30 eyes that will be treated with external DCR with anastomosis of posterior mucosal flaps .

Group B: includes 30 eyes that will be treated with external DCR with amputation of posterior mucosal flaps .

Study Population:

Study participants will be: 60 eyes undergo external DCR . All patients included in this study will be verbally briefed about the details and the nature of the study & will sign a written consent according to the local Ethics Committee of Minia University Faculty of Medicine. The study will be conducted in Ophthalmology department, Minia university Hospital, Egypt.

ELIGIBILITY:
Inclusion criteria

* Patients with chronic dacryocystits,
* primary nasolacrimal duct obstruction
* Lacrimal mucocele
* Lacrimal fistula

Exclusion Criteria:

* Recurrent cases.
* Age under 5 years.
* Associated nasal pathology.
* Sever dry eye
* Patients unfit for general anaesthesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Management of posterior flap in external DCR | patient evaluated at 2 months after surgery then at 4th month then 6th month
  Evaluation of different methods of posterior flaps management in external dacryocystorhinostomy using nasal endoscopy for evaluation of outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine ,Minia university, Minya, Egypt